CLINICAL TRIAL: NCT03318562
Title: A Pharmacodynamic Study of Oral eFT508 in Subjects With Advanced Triple Negative Breast Cancer and Hepatocellular Carcinoma
Brief Title: A PD Study of Oral eFT508 in Subjects With Advanced TNBC and HCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to change in focus of the development program
Sponsor: Effector Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eFT508-0008
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2017-12

CONDITIONS: Triple Negative Breast Cancer; Hepatocellular Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Hepatocellular | interventions — tomivosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNBC Cohort (Experimental): female subjects who have pathologically documented, radiographically measurable, metastatic or locally advanced and unresectable TNBC and have received >=1 prior cancer therapy regimen for metastatic disease
  Interventions: Drug: eFT508
- HCC Cohort (Experimental): male and female subjects who have histologically or cytologically confirmed advanced HCC not amenable to surgical resection and have failed >=1 systemic therapy, which must include sorafenib, or are intolerant to multikinase inhibitor therapies
  Interventions: Drug: eFT508

INTERVENTIONS:
Drug: eFT508 — 200 mg eFT508 dosed BID for 3 week cycles

SUMMARY:
This study will evaluate the pharmacodynamic (PD), safety, antitumor activity, and PK of eFT508 in female subjects who have pathologically documented, radiographically measurable, metastatic or locally advanced and unresectable TNBC and have received prior cancer therapy regimen for metastatic disease, and in male and female subjects who have histologically or cytologically confirmed advanced HCC not amenable to surgical resection and have failed systemic therapy.

ELIGIBILITY:
Inclusion Criteria (TNBC Cohort Only):

* Women ≥18 years of age
* Pathologically documented diagnosis of TNBC that is metastatic or locally advanced and unresectable
* Adequate hepatic function and coagulation profile
* Negative HIV, HBV and HCV

Inclusion Criteria (HCC Cohort Only):

* Men or Women ≥18 years of age
* Histological or cytological confirmed diagnosis of HCC with Barcelona Clinic Liver Cancer Stage B or C who cannot benefit from resection, local ablation, or chemoembolization
* ECOG performance status of 0 or 1
* Has at least 1 measurable lesion based on irRECIST 1.1.
* Negative HIV tests

Inclusion Criteria (Either Cohort):

* subject agrees to undergo a pre-treatment and an on-treatment biopsy of the tumor
* Completion of all previous therapy for the treatment of cancer ≥3 weeks before the start of study drug
* All acute toxic effects of any prior antitumor therapy resolved to Grade ≤1 before the start of study drug
* Adequate bone marrow and renal function
* Life expectancy of ≥3 months

Exclusion Criteria (Either Cohort):

* Pregnant or breastfeeding
* History of another malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin; in situ cervical carcinoma; adequately treated, papillary, noninvasive bladder cancer; other adequately treated Stage 1 or 2 cancers currently in complete remission; or any other cancer that has been in complete remission for ≥2 years.
* Gastrointestinal disease that may interfere with drug absorption or with interpretation of GI AEs.
* Known symptomatic brain metastases requiring ≥10 mg/day of prednisolone (or its equivalent).
* Significant cardiovascular disease within 6 months prior to start of study drug
* Ongoing risk for bleeding due to active peptic ulcer disease or bleeding diathesis or requirement for systemic anticoagulation with unfractionated heparin, low-molecular-weight heparin or heparin fractions, or oral anticoagulants.
* Evidence of an ongoing systemic bacterial, fungal, or viral infection
* Has received a live vaccine within 30 days of planned start of study drug
* Major surgery within 4 weeks before the start of study drug
* Prior solid organ or bone marrow progenitor cell transplantation
* Prior therapy with any known inhibitor of MNK1 or MNK2
* Prior high dose chemotherapy requiring stem cell rescue
* History of or active autoimmune disorders or other conditions that might impair or compromise the immune system
* Ongoing immunosuppressive therapy, including systemic or enteric corticosteroids
* Use of a strong inhibitor or inducer of cytochrome P450 (CYP)3A4 within 7 days prior to the start of study drug or expected requirement for use of a strong CYP3A4 inhibitor or inducer during study participation
* Need for proton pump inhibitors and histamine H2 blockers
* Previously received investigational product in a clinical trial within 30 days or within 5 elimination half lives (whichever is longer) prior to the start of study drug, or is planning to take part in another clinical trial while participating in this study
* HCC Cohort Only: Portal vein invasion at the main portal (Vp4), inferior vena cava, or cardiac involvement of HCC based on imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Level of biomarkers of antitumor activation | 28 days
  Biomarkers of antitumor immune activation in pre- and on treatment tumor biopsies and peripheral blood cells

SECONDARY OUTCOMES:
Molecular profiling of circulating lymphocytes and tumor-infiltrating lymphocytes (TILs) | up to 3 years
  Includes determination of T cell clonality via T cell receptor sequencing
Levels of eIF4E and phospho-eIF4E | up to 3 years
  Assessment of eIF4E and phospho-eIF4E in tumor biopsies by immunohistochemistry, and in circulating peripheral blood cells by phospho-flow cytometry
Number of mutations | up to 3 years
  Assessment of mutations will be determined for a subset of known cancer driver genes by sequencing tumor DNA
Objective tumor response | up to 3 years
  determined by irRECIST 1.1, defined as the proportion of subjects who achieve a complete response (CR) or partial response (PR)
Progression Free Survival | up to 3 years
  as determined by irRECIST 1.1, defined as the interval from the start of study drug to the earlier of the first documentation of disease progression or death from any cause
Proportion of subjects with TEAEs and SAEs | up to 3 years
PK plasma concentrations | up to 21 weeks
  taken at the anticipated maximum and minimum plasma concentrations for eFT508

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Barton, MD, Study Director — CMO
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Kansas City Research Institute, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No